CLINICAL TRIAL: NCT07062107
Title: Study on the Application of Adaptive Fluidics Technique in the Surgery of Lens Diseases
Brief Title: Study on the Application of Adaptive Fluidics Technology in Lens Diseases Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-0063
Record Dates: First submitted 2025-06-24; First posted 2025-07-14 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-06

CONDITIONS: Lens Diseases
MeSH Terms: conditions — Lens Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional fluidics for phacoemulsification (Active Comparator): Traditional fluidics systems are used for perfusion during phacoemulsification.
  Interventions: Procedure: Conventional phacoemulsification surgery
- Adaptive fluidics for phacoemulsification (Experimental): Adaptive fluidics technology are used for perfusion during phacoemulsification.
  Interventions: Procedure: Phacoemulsification using adaptive fluidics technology

INTERVENTIONS:
Procedure: Conventional phacoemulsification surgery — Conventional phacoemulsification surgery adopts the traditional perfusion system and uses intraoperative optical coherence tomography to assist in observation.
  Other Names: Phacoemulsification using traditional fluidics
  Arms: Traditional fluidics for phacoemulsification
Procedure: Phacoemulsification using adaptive fluidics technology — Phacoemulsification surgery adopts the adaptive fluidics system to precisely and dynamically control the pressure and flow rate of the perfusion fluid. During the operation, optical coherence tomography is used to assist in observing the stability of the anterior chamber.
  Other Names: Phacoemulsification using adaptive fluidics
  Arms: Adaptive fluidics for phacoemulsification

SUMMARY:
In phacoemulsification surgery for lens diseases using a traditional fluidics technology with a fixed perfusion pressure, the moment the perfusion needle enters the anterior chamber, the intraocular pressure will increase sharply. Moreover, the perfusion pressure cannot change along with the intraocular pressure during the operation, giving rise to many risks and threatening the safety of the surgery. The aim of this study is to apply adaptive fluidics technology to dynamically and precisely regulate the pressure and flow rate of the perfusion fluid, maintaining a relatively stable intraocular pressure during the operation. Meanwhile, intraoperative optical coherence tomography（OCT）was utilized to assist in observing the intraocular conditions, to study the advantages of adaptive fluidics technology in maintaining anterior chamber stability, and to verify the clinical application value of this technology in different types of lens diseases.

DETAILED DESCRIPTION:
Phacoemulsification is currently the most commonly used surgical method for lens diseases. During the operation, it is necessary to continuously deliver perfusion fluids such as balanced salt solution into the eye (anterior chamber) to maintain the depth of the anterior chamber and the stability of intraocular pressure. The perfusion pressure of the traditional fluidics system is constant, which may lead to problems such as a sudden increase in intraocular pressure at the moment the perfusion needle enters the eye, thereby increasing the surgical risk and affecting the surgical outcome. How to ensure that the intraocular pressure of patients remains relatively stable during surgery, optimize the surgical process and achieve a better prognosis has received extensive attention from ophthalmology practitioners and researchers. The emergence and application of adaptive fluidics can dynamically optimize the pressure and flow rate of perfusion fluid during surgery, significantly reduce intraocular pressure fluctuations, and enhance the stability of the anterior chamber. At present, the relevant research on the application of adaptive fluid flow technology to assist in lens disease surgery is still scarce. Its exact application value and practical advantages still need to be fully verified and elaborated in detail through clinical trials, follow-up observations and other links. The aim of this study is to apply adaptive fluidics technology to dynamically and precisely regulate the pressure and flow rate of the perfusion fluid, maintaining a relatively stable intraocular pressure during the operation. Meanwhile, intraoperative optical coherence tomography（OCT）was utilized to assist in observing the intraocular conditions, to study the advantages of adaptive fluidics technology in maintaining anterior chamber stability, and to verify the clinical application value of this technology in different types of lens diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lens opacity or abnormal position, with or without anterior segment structural changes, who meet the surgical indications and are aged between 18 and 80 years old and require lens surgery.

Exclusion Criteria:

* The patient has severe corneal scars or other corneal lesions, intraocular inflammation, and lesions of the retina, choroid, optic nerve, etc. that seriously affect the prognosis of vision. The patient has a clear history of systemic diseases affecting vision, a history of systemic medication, concurrent retinopathy, and other contraindications for conventional lens surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Real-time intraocular pressure changes during the operation | During the operation
  The variation range of intraocular pressure during phacoemulsification surgery, especially the intraocular pressure at the moment when the perfusion needle enters the anterior chamber.
Quantify the measured values of ultrasonic energy exposure | During the operation
  Including average phacoemulsification energy, average phacoemulsification power, effective phacoemulsification time and total phacoemulsification time.
The volume of perfusion fluid used during the operation | During the operation
  Including average perfusion time, average aspiration time, average flow rate and total liquid usage.
Intraoperative OCT-assisted observation of anterior chamber depth changes | During the operation
  Using intraoperative OCT to evaluate the distance between the pupil margin and the corneal endothelium to measure the changes in anterior chamber depth.

SECONDARY OUTCOMES:
Technical indicators related to anterior segment OCT during the operation | During the operative
  Using intraoperative OCT to record the technical indicators related to the anterior segment.
Intraocular pressure | 1day, 1 week, 1 month and 3 month postoperation
Successful implantation rate of intraocular lens | Through study completion, an average of 1 year
  Implantation rate of intraocular lens after surgery
Intraocular lens position after implantation | 1day, 1 week and 1 month postoperation
  The location of intraocular lens after surgery, observed through slit - lamp and anterior segment optical coherence tomography.
Visual function | 1day, 1 week, 1 month and 3month postoperation
  Best corrected visual acuity (BCVA) measured using a decimal chart Best corrected visual acuity (BCVA) measured using a decimal chart
Postoperative complication | 1 week, 1 month and 3month postoperation

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine,, Hangzhou, Zhejiang, China